CLINICAL TRIAL: NCT00051623
Title: A Multicenter, Randomized, Double-blind Trial of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab) for the Treatment of Patients With Psoriatic Arthritis
Brief Title: A Study of the Safety and Effectiveness of Infliximab for the Treatment of Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004789
Record Dates: First submitted 2003-01-14; First posted 2003-01-15 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic arthritis; Infliximab; Remicade
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to determine if Infliximab is safe and effective in the treatment of psoriatic arthritis. Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce painful disease.

DETAILED DESCRIPTION:
This is a phase III, multicenter, randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled study designed to determine the safety and effectiveness of Infliximab in the treatment of patients with psoriatic arthritis. This is an experimental medical research study. A total of 200 people in North America and Europe participated in this study during the 17 month study period. Patients will receive infusions of either placebo or 5 or 10 mg/kg infliximab (Remicade) at weeks 0,2, 6, 14, 16, 18, 22, 30, 38, and 46. Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive either placebo or 5 mg/kg induction infusions (weeks 0, 2 and 6) followed by maintenance infusions every 8 weeks until week 46. In the placebo group, patients may early escape at week 16 and crossover at week 24 to infliximab;. In the 5mg/kg group, dose escalation if needed at week 38.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed psoriatic arthritis for >= 6 months
* active arthritis with >= 5 tender and 5 swollen joints
* active psoriasis

Exclusion Criteria:

* Have other inflammatory diseases, including but not limited to, rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, or Lyme disease
* Received any systemic immunosuppressives within 4 weeks prior to enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-05; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with American College of Rheumatology (ACR) 20 response at week 14 Change from baseline in total radiographic scores of hands and feet at week 24

SECONDARY OUTCOMES:
Number of patients who achieved an ACR 20 response at wk 24; PsARC at wk 14; proportion of patients with >= to 75% Improvement From Baseline in PASI at Week 14; change from baseline SF 36 physical component summary scores at wk 14

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Background] Bortul M, Calligaris L, Moro E, Bazzocchi M, Strami G. [Preoperative transhepatic biliary drainage in the jaundiced patient: our experience]. Ann Ital Chir. 1991 May-Jun;62(3):265-71; discussion 272. Italian. PMID 1755609
- [Result] Kavanaugh A, Antoni C, Mease P, Gladman D, Yan S, Bala M, Zhou B, Dooley LT, Beutler A, Guzzo C, Krueger GG. Effect of infliximab therapy on employment, time lost from work, and productivity in patients with psoriatic arthritis. J Rheumatol. 2006 Nov;33(11):2254-9. Epub 2006 Sep 1. PMID 16960923
- [Result] Kavanaugh A, Krueger GG, Beutler A, Guzzo C, Zhou B, Dooley LT, Mease PJ, Gladman DD, de Vlam K, Geusens PP, Birbara C, Halter DG, Antoni C; IMPACT 2 Study Group. Infliximab maintains a high degree of clinical response in patients with active psoriatic arthritis through 1 year of treatment: results from the IMPACT 2 trial. Ann Rheum Dis. 2007 Apr;66(4):498-505. doi: 10.1136/ard.2006.058339. Epub 2006 Nov 17. PMID 17114188
- [Result] van der Heijde D, Kavanaugh A, Gladman DD, Antoni C, Krueger GG, Guzzo C, Zhou B, Dooley LT, de Vlam K, Geusens P, Birbara C, Halter D, Beutler A. Infliximab inhibits progression of radiographic damage in patients with active psoriatic arthritis through one year of treatment: Results from the induction and maintenance psoriatic arthritis clinical trial 2. Arthritis Rheum. 2007 Aug;56(8):2698-707. doi: 10.1002/art.22805. PMID 17665424
- [Derived] Englbrecht M, Wang Y, Ronneberger M, Manger B, Vastesaeger N, Veale DJ, Schett G. Measuring joint involvement in polyarticular psoriatic arthritis: an introduction of alternatives. Arthritis Care Res (Hoboken). 2010 Jul;62(7):977-83. doi: 10.1002/acr.20161. PMID 20191568
- See also: A Multicenter, Randomized, Double-blind Trial of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab) for the Treatment of Subjects with Psoriatic Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=153&filename=CR004789_CSR.pdf
- See also: |A Multicenter, Randomized, Double-blind Trial of Anti TNFa Chimeric Monoclonal Antibody (Infliximab) for the Treatment of Subjects with Psoriatic Arthriti — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=153&filename=CR004789_REF1.pdf